CLINICAL TRIAL: NCT03386968
Title: Use of Low-Cost Virtual Reality and Active Video Games to Improve Balance and Perceptual Skills in Children With Cerebral Palsy and Brain Injury
Brief Title: Virtual Reality and Active Video Games to Improve Balance in Children With Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blythedale Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-1206TS
Record Dates: First submitted 2017-12-07; First posted 2017-12-29 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy; Acquired Brain Injury
Keywords: virtual reality; hemiplegia; diplegia; video gaming; active video games; Playstation X-Box 360; Rutgers V-Step; Microsoft Kinect
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries; Hemiplegia | interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: A Randomized Block Design will be utilized in order to attempt to "match" subjects according to functional level and diagnosis (cerebral palsy or acquired brain injury). Upon signing consent the subjects will be grouped based on their diagnosis. At that time gait speed for the 10 M Walk Test will be utilized to categorize all participants into a "fast" and "slow" group. (subjects performing the 10 M Walk Test at a speed less than .4 m/s will be placed in the "slow" group, and subjects testing at a speed greater than or equal to .4 m/s will be placed in the "fast" group After this determination is made, subjects will be randomized to "control" (usual care), and "intervention" one therapy session replaced with a session utilizing Active video games and the Rutger's V-step. A minimum of 2 subjects per grouping will be sought in order to analyze for differences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video gaming (Experimental): A child's usual physical therapy session will be replaced with a session utilizing Active video games and the Rutger's V-step.
  Interventions: Behavioral: Active video gaming
- Usual care (Active Comparator): Children will receive their usual care in the physical therapy program at Blythedale.
  Interventions: Behavioral: Usual care physical therapy

INTERVENTIONS:
Behavioral: Active video gaming — Children will visit Blythedale for 8 sessions, one 45-session visit per week, in place of one of the child's typical physical therapy sessions. During each session, children will play a video game on the X-Box Kinect system, using the games "Kinect Adventures" and "Kinect Sports". The child will first play a "Kinect Adventures" game, which requires ambulating, ducking, and dodging one's way through an obstacle course.
  Arms: Video gaming
Behavioral: Usual care physical therapy — Children will attend their usual care physical therapy appointments at Blythedale.
  Arms: Usual care

SUMMARY:
The purpose of this pilot feasibility study is to assess the feasibility of using the Playstation Xbox 360 and Rutgers V-step via a Kinect Sensor with active video game software as a part of a physical therapy intervention to improve obstacle negotiation, gait speed, and stair negotiation in ambulatory children with Cerebral Palsy (CP) hemiparesis or spastic diplegia, or non-progressive brain injury (BI). Children will be assessed using perceptual, balance, functional and gait assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-17
* Diagnosis of Cerebral Palsy or Diagnosis of Acquired Brain Injury
* Ambulatory with or without an assistive device x 150 feet
* Cognition and attention ability sufficient to be successful in video game play and to follow instructions of the investigator.
* Able to complete testing process.
* Current patient at Blythedale Children's Hospital program (Expected Length of Stay/availability for study of approximately 8 weeks)

Exclusion Criteria:

* Any history of photosensitive epilepsy or seizures triggered by exposure to flashing lights, television or video games
* Attention or behavior problems that prevent the successful completion of game play
* Any acute musculoskeletal injury that limits weight bearing on one lower extremity (due to orthopedist concerns for fracture or injury)
* Any medical condition that prevents the child from tolerating exercise due to cardiovascular conditions

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Change in Pediatric Evaluation of Disability Inventory Computer Adaptive Test | From before intervention to immediately after intervention
  The PEDI-CAT measures abilities in three functional domains: Daily Activities, Mobility and Social/Cognitive.

SECONDARY OUTCOMES:
Change in 10 Meter walk test | From before intervention to immediately after intervention
  Measures time taken for a participant to walk 10 meters
Change in Gross Motor Function Measure (GMFM) subtest D and E | From before intervention to immediately after intervention
  The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy.
Change in Four Square Step Test | From before intervention to immediately after intervention
  Measures how well a patient can change directions while stepping.
Change in Functional Gait Assessment (FGA) | From before intervention to immediately after intervention
  10-item test that assesses dynamic balance and postural stability during gait.
Change in Motor Free Visual Perceptual Test (MVPT)-4 | From before intervention to immediately after intervention
  The MVPT-4 assesses five categories of visual perception: Visual Discrimination: Ability to discriminate dominant features of different objects, including the ability to discriminate position, shapes, and forms.
Change in Visually guided weight shift ability as measured by the Smart Balance Master® | From before intervention to immediately after intervention
  Force platform system that tests balance
Change in Children's Assessment of Participation and Enjoyment | From before intervention to immediately after intervention
  Self-report measures of children's participation in recreation and leisure activities outside of mandated school activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Blythedale Children's Hospital, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: No